CLINICAL TRIAL: NCT01223079
Title: Use of r-hLH (Luveris) Late Follicular Phase for Controlled Ovarian Stimulation (COS) in Donor Patients Previously Treated With r-hFSH (Gonal F)in a Long Luteal Downregulated Cycle With GnRH Agonist. A Cross-over Study
Brief Title: Use of r-hLH (Luveris) in Donors Previously Treated With r-hFSH (Gonal F)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20052361
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Outcome During r-hFSH Stimulation; Outcome During r-hFSH and r-hLH Stimulation
Keywords: r-hFSH; r-hLH
MeSH Terms: interventions — follitropin alfa; Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- r-hFSH (Gonal F) (Other): Patients will be treated with r-hFSH throughout the stimulation phase of their first cycle until r-hCG administration.
  Interventions: Drug: r-hFSH
- r-hFSH (Gonal F) and r-hLH (Luveris) (Other): Patients will be treated with r-hFSH only until they have 2 follicles greater than or equal to 14mm. Patients will then bring 300IU/day of r-hLH until r-hCG administration.
  Interventions: Drug: r-hFSH and r-hLH

INTERVENTIONS:
Drug: r-hFSH — r-hFSH dose to be determined by the patient's primary doctor and adjusted according to their response
  Other Names: Gonal F
  Arms: r-hFSH (Gonal F)
Drug: r-hFSH and r-hLH — Patients will begin r-hLH at 300IU/day when there are 2 follicles greater than or equal to 14mm.
  Other Names: r-hFSH; Gonal F; r-hLH; Luveris
  Arms: r-hFSH (Gonal F) and r-hLH (Luveris)

SUMMARY:
The purpose of the study is to compare the safety and efficacy of r-hLH to r-hFSH in the late follicular phase of young women undergoing controlled ovarian stimulation for oocyte donation.

DETAILED DESCRIPTION:
While the role of FSH is considered the fundamental driver of folliculogenesis, the role of LH in this process is more controversial. FSH is associated with stimulating growth and recruitment of follicles while LH is associated with the selection of dominant follicles destined for ovulation. We will use an open, prospective, cross-over study to compare the safety and efficacy of two different treatment protocols for controlled ovarian stimulation in egg donors.

20 participants will undergo two cycles of stimulation. The first one will be with r-hFSH though the cycle and the second with r-hFSH then r-hLH. The participants will have 1 month rest cycle between the treatment cycles. r-hFSH doses will be adjusted according to patient response. r-hLH dosing will begin when there are 2 follicles greater than or equal to 14mm in diameter. The does will be 300IU/day and continue until the day of r-hCG administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than or equal to 32 years old
2. BMI<35
3. Eligible for controlled ovarian simulation
4. No PCO-type ovaries (PCO by USS image, >2.1 LH;FSH ratio on cycle day 3, insulin resistance, increase of testosterone over free testosterone)
5. Meet all requirements for becoming an egg donor
6. Willingness and ability to participate and comply with study protocol for the duration of the study
7. Baseline FSH<11

Exclusion Criteria:

1. Clinically significant systemic disease
2. Any contraindication to gonadotropin therapy
3. LH:FSH ratio greater than 3
4. Pregnancy in the past 3 months
5. Any medical condition which, in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug
6. Simultaneous participation in another clinical trial
7. Known active substance abuse, including tobacco and alcohol (>10 cigarettes/day)
8. Refusal or inability to comply with protocol
9. Known poor ovarian response

Ages: 21 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of r-hFSH protocol | 6 months
  Evaluation of the safety and efficacy of r-hFSH for controlled ovarian stimulation in the same patients.
Safety and efficacy of r-hFSH + r-hLH protocol | 6 months
  Evaluation of the safety and efficacy of r-hFSH for controlled ovarian stimulation in the same patients.

SECONDARY OUTCOMES:
Number of oocytes retrieved | 6 months
  Evaluation of the number of oocytes obtained as a function of stimulation protocol.
Quality of embryos obtained | 6 months
  Evaluation of pregnancy rates (clinical and ongoing), delivery rates, multiple pregnancy rates and the number of cancelled cycles.
Incidences of ovarian hyperstimulation syndrome | 6 months
  Evaluation of the potential adverse effects associated with ovarian stimulation
Quality of oocytes obtained | 6 months
  Evaluation of the quality of oocytes obtained as a function of stimulation protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Morristown, New Jersey, United States